CLINICAL TRIAL: NCT02213081
Title: Phase IV Pilot Study of Ulipristal Acetate for Treatment of Endometriosis-related Pelvic Pain
Brief Title: Ulipristal for Endometriosis-related Pelvic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00091840
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Endometriosis
Keywords: Endometriosis; chronic pelvic pain; dysmenorrhea; dyschezia; bleeding; ulipristal; progesterone
MeSH Terms: conditions — Endometriosis; Dysmenorrhea; Constipation; Hemorrhage | interventions — ulipristal; ulipristal acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ulipristal (Experimental): 1 patient with chronic, endometriosis-related pelvic pain refractory to medical and/or surgical therapies will receive 15mg ulipristal every other day (three times a week- Monday, Thursday, Saturday) for three months.
  Interventions: Drug: Ulipristal

INTERVENTIONS:
Drug: Ulipristal — Patient will take 15mg every other day, or every 4 days per week.
  Other Names: Ulipristal Acetate; Ella

SUMMARY:
The aim of this research is to assess the benefit of a medication (ulipristal) for alleviation of symptoms in women with chronic, endometriosis-related pelvic pain.

DETAILED DESCRIPTION:
This study will assess the use of a medication to improve symptoms of chronic, endometriosis-related pelvic pain among women who did no achieve relief with prior surgical and medical treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of endometriosis with surgical confirmation via laparoscopy performed within 3 years prior to study enrollment
* English-speaking reproductive-age women (18-50yo) with regular, cyclical menses
* Treatment-refractory endometriosis, as defined by persistent or recurrent pelvic pain following one or more treatments involving surgery and/or hormonal treatment
* Dysmenorrhea and chronic pelvic pain for a least one week out of the month during past 5 months or longer
* Endometrial biopsy before and after intervention
* Adequate organ and marrow function as defined below:
* leukocytes ≥ 3,000/microliter
* absolute neutrophil count ≥ 1,500/microliter
* platelets ≥ 100,000/microliter
* total bilirubin within normal institutional limits
* Liver function tests ≤ 2.5 X institutional upper limit of normal
* creatinine within normal institutional limits
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Undiagnosed vaginal bleeding
* Abnormal results from endometrial biopsy
* Presence of ovarian cysts ≥ 3 cm
* Pregnancy
* Refusal to adhere the birth control strategy of the study (use of a combination of a condom and a vaginal sponge during each intercourse while on ulipristal, plus one month before the onset and one month after the completion of ulipristal therapy)
* Women taking digoxin, dabigatran or etexilate due to interference of ulipristal acetate with the concentration of these substances bound by plasma proteins.
* Women taking moderate to potent inducers of hepatic metabolism (e.g. erythromycin, ketoconazole, ritonavir, nefazodone).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Ulipristal.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active pulmonary, cardiac, renal, hepatic or thromboembolic disease, infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Bulun, Principal Investigator — Northwestern University, Northwestern Memorial Hopsital
Locations (1):
- Northwestern University, Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ulipristal: 1 patient with chronic, endometriosis-related pelvic pain refractory to medical and/or surgical therapies received 15mg ulipristal every other day (three times a week- Monday, Thursday, Saturday) for three months.
Period: Overall Study
Arm/Group | Ulipristal
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ulipristal
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 25 [25 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Pelvic Pain
Description: Scores were collected daily and averaged together for each period
Time Frame: Patients will document self-reported daily pain scores via visual analogue scale(0 to10 where 0 is no pain and 10 is worst pain)for one month prior to starting treatment (1 month),while receiving treatment (3 months) after cessation of treatment (1 month)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ulipristal
Number analyzed (Participants) | 1
units on a scale
  Prior to starting therapy | 3.5 (0.57)
  During therapy | 0.2 (0.06)
  After cessation of therapy | 3.9 (0.43)
Statistical Analysis 1: Comparison: Ulipristal; Test type: Equivalence — Wilcoxon signed rank test was used to determine if the mean difference in pain scores before compared to during ulipristal therapy were equivalent or non-equivalent; p < 0.05, Wilcoxon signed rank; Mean Difference (Net) = 3.5, Standard Error of Mean 0.57

2. Secondary Outcome: Vaginal Bleeding
Description: Patient will record the # of tampons or pads they use each week while enrolled in the study (1 month pre-medication, 3 months during medication, 1 month after medication).
Time Frame: 5 months
Measure: Number; unit: pads or tampons
Arm/Group | Ulipristal
Number analyzed (Participants) | 1
pads or tampons
  Prior to therapy | 3
  During therapy | 0
  After cessation of therapy | 3

3. Secondary Outcome: Pain With Sexual Intercourse
Description: If sexually active, patients will document self-reported weekly average pelvic pain scores (0 to 10 where 0 is no pain and 10 is worst pain) with sexual intercourse for one month prior to starting treatment, while receiving treatment for 3 months and for one full month subsequent to treatment.
Time Frame: 5 months
Population: The one patient in our study was not sexually active during her enrollment in the study such that dyspareunia pain scores were unable to be assessed.
Arm/Group | Ulipristal
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Pain With Bowel Movements
Description: Patient will document self-reported weekly average pelvic pain scores with defecation (0 to 10 where 0 is no pain and 10 is worst pain) for one month prior to starting treatment, while receiving treatment for 3 months and for one full month subsequent to treatment.
Time Frame: Patient will document self-reported daily pain scores via visual analogue scale(0 to 10 where 0 is no pain and 10 is worst pain) for one month prior to starting treatment (1 month),while receiving treatment (3 months)after cessation of treatment(1 month)
Population: Our one patient did not report dyschezia before, during, or after ulipristal treatment.
Measure: Number; unit: units on a scale
Arm/Group | Ulipristal
Number analyzed (Participants) | 1
units on a scale
  Prior to treatment | 0
  During treatment | 0
  After treatment | 0

ADVERSE EVENTS:
Arm/Group | Ulipristal
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No